CLINICAL TRIAL: NCT01585311
Title: Impact of Prolonged Tachycardia on Cardiovascular Morbidity and Outcome After Subarachnoid Hemorrhage (SAH)
Brief Title: Impact of Tachycardia on Outcome After Subarachnoid Hemorrhage (SAH)
Status: Terminated | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: AAAA5384
Record Dates: First submitted 2012-04-24; First posted 2012-04-25 (Estimated); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Subarachnoid Hemorrhage (SAH); Tachycardia
Keywords: Subarachnoid Hemorrhage (SAH); tachycardia; Outcome
MeSH Terms: conditions — Subarachnoid Hemorrhage; Tachycardia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subarachnoid Hemorrhage patients: SAH patients with hourly eMR values of Heart Rate

SUMMARY:
The purpose of this retrospective study is to test the hypothesis that uncontrolled tachycardia serves as a risk factor for adverse cardiovascular events and poor outcome after Subarachnoid Hemorrhage (SAH).

DETAILED DESCRIPTION:
The design of the current study will be to conduct a retrospective analysis of prolonged heart rate and uncontrolled tachycardia using patients enrolled in the investigators prospective observational cohort study since the electronic medical record systems have been implemented. The investigators know that there have been periods when these electronic systems have failed, resulting in lost data. The investigators anticipate retrospective collection of hourly heart rate for approximately 400 SAH patients that will have ICU data and 3 month modified Rankin documented in our Subarachnoid Hemorrhage Outcomes Project (SHOP) database. The investigators will determine what percent of them have prolonged elevated heart rate and tachycardia. Prolonged heart rate and uncontrolled tachycardia has been defined as a heart rate greater than 95 for greater than 12 hours in one 24 hour period of their ICU stay. The investigators will conduct a ROC curve analysis to determine the appropriate heart rate and duration thresholds that are most predictive of poor prognosis after SAH. Patients be will stratified based on several criteria including admission coma score, early (SAH day 0 to 3) or late (SAH day >=4) ICU admission, presence of intraventricular hemorrhage on admission CT, history of beta-blocker usage, age, and gender.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 years
* Diagnosis of subarachnoid hemorrhage established by computed tomography (CT scan) or xanthochromia of the cerebrospinal fluid if the CT is negative
* Written informed consent from either the patient or a family member
* Admitted to the NICU for at least 12 hours

Exclusion Criteria:

* Age < 18yrs
* traumatic SAH
* SAH due to a rupture of an arteriovenous malformation, neoplasm vasculitis or other secondary causes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the Columbia Neurocritical Care Unit with a diagnosis of subarachnoid hemorrhage established by computed tomography (CT scan) or xanthochromia of the cerebrospinal fluid if the CT is negative.
Sampling Method: Non-Probability Sample
Enrollment: 1540 (Actual)
Dates: Start 2008-03; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
modified Rankin Scale (mRS) score | Three months

SECONDARY OUTCOMES:
Prevalence of Major Adverse Cardiovascular Events (MACE) | 3 months
  1. pulmonary edema,
  2. severe hypertension or
  3. hypotension requiring IV infusion therapy,
  4. myocardial infarction, and
  5. serious cardiac arrhythmias including sudden cardiac arrest.
  6. length of ICU and hospital stay for patients with and without uncontrolled tachycardia

CONTACTS AND LOCATIONS:
Overall Officials: Jan Claassen, MD, Principal Investigator — Columbia University; J. Michael Schmidt, PhD, Study Director — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States